CLINICAL TRIAL: NCT01856608
Title: Assessing the Utility of the Team SA Instrument in Measuring the Effectiveness of Communication Across Disciplines During ICU Rounds
Brief Title: Assessing the Team SA Instrument in Measuring the Effectiveness of Communication Across Disciplines During ICU Rounds
Status: Completed | Type: Observational
Sponsor: Naeem Ali, MD (Other)
Responsible Party: Sponsor-Investigator, Naeem Ali, MD, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2012B0233
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2013-07

CONDITIONS: Personal Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Assessing the utility of the Team SA instrument in measuring the effectiveness of communication across disciplines during ICU rounds.

DETAILED DESCRIPTION:
Multidisciplinary rounds are events that occur daily in Intensive care units. During these events, practitioners from multiple disciplines meet at a pre-specified time to discuss current medical condition and plans of care. At the conclusion of these discussions, all practitioners are expected to understand the plan of care well enough to execute defined tasks, but also coordinate as circumstances change. In order to coordinate under changing circumstances practitioners must have a broader understanding of the current state of the patient and how likely certain deteriorations are. This synthetic understanding of patient risks across multi-provider groups has been described as anticipatory team situational awareness (Team SA). One instrument has been validated in the ICU as feasible and informative. This Team SA survey successfully identified that the time spent in "training" discussions improved Team SA across physician groups. The investigators' goal is to implement this survey across the investigators' medical ICU service to obtain a baseline estimate of how effective current communication patterns are for achieving concordant Team SA. If gaps in communication are encountered future interventions will be developed

ELIGIBILITY:
Inclusion Criteria:

* Nurses, primary clinicians (resident or NP) and Critical Care physicians (Staff or Fellow in Critical Care Medicine) will be approached for interview. All subjects will be approached individually and asked to participate outside of the presence of the other potential study subjects.

Exclusion Criteria:

* N/A

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Daily census rosters of the MICU and 8ICU nursing units will be reviewed for occupancy. At 8am on survey days occupied beds will be tallied (up to 39 beds). Beds occupied by a non-MICU service patient and those with active DNR-CC orders will be excluded. From the remaining patients, ten bed numbers will be randomly selected for review. Randomization will be stratified by MICU service sub-unit (MICU 40, MICU 90, 8ICU). If fewer than ten patients are eligible on an assigned survey day, all patients in the ICU on that day will be surveyed.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To determine if it is feasible to survey clinicians regarding their opinions about future risks for individual patients in the ICU setting To determine the range of team situational awareness exhibited by current ICU clinician teams | It is expected that a maximum of ten minutes will be required to complete the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Ali, MD, Principal Investigator — Ohio State University
Locations (1):
- Davis Heart and Lung Research Institute 473 w. 12TH aVE, Columbus, Ohio, United States